CLINICAL TRIAL: NCT02019706
Title: Prospective Evaluation of 68Ga-DOTATATE PET/CT, Octreotide and F-DOPA PET Imaging in Ectopic Cushing Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140028; 14-CH-0028
Record Dates: First submitted 2013-12-21; First posted 2013-12-24 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-04-09

CONDITIONS: ACTH; Cushing's Syndrome
Keywords: DOTATATE; Cushing's Syndrome; Hypercortisolism
MeSH Terms: conditions — Cushing Syndrome | interventions — gallium Ga 68 dotatate; fluorodopa F 18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imaging (Experimental): All subjects will be imaged
  Interventions: Radiation: DOTATATE PET-CT; Radiation: F-DOPA PET CT; Radiation: CT scan; Diagnostic Test: Routine MRI scan; Diagnostic Test: Gated MRI scan; Drug: 68Ga-DOTATATE; Drug: 18F-DOPA

INTERVENTIONS:
Radiation: DOTATATE PET-CT — 68Ga-DOTATATE PET/CT
Radiation: F-DOPA PET CT — 68Ga-DOTATATE PET/CT
Radiation: CT scan — routine CT scan
Diagnostic Test: Routine MRI scan — routine 1.5 or 3T MRI scan
Diagnostic Test: Gated MRI scan — Cardiac gated MRI scan
Drug: 68Ga-DOTATATE — 68Ga-DOTATATE radioligand
Drug: 18F-DOPA — 18F-DOPA radioligand

SUMMARY:
Between 10% and 15% of patients with endogenous hypercortisolism (Cushing syndrome) have ectopic (non-pituitary) production of adrenocorticotropin hormone (ACTH) that causes cortisol excess. In approximately 50% of these patients, the tumoral source of ACTH cannot be found initially despite very detailed and extensive imaging, including studies such as computed tomography, magnetic resonance imaging, and octreotide scan (Octreoscan) using the standard dose of indium- 111 pentetreotide ([111In-DTPA-D-Phe]-pentetreotide). The sensitivity and specificity of structurally based imaging studies depends on anatomic alterations and the size of the tumor. In contrast, positron emission tomography (PET) and somatostatin ligand imaging detect pathologic tissue based on physiologic and biochemical processes within the abnormal tissue. This protocol tests the ability of [18F]-L-3,4-dihydroxyphenylalanine (18F-DOPA) PET, and the somatostatin imaging analogue, 68Ga-DOTATATE-PET, to localize the source of ectopic ACTH production.

...

DETAILED DESCRIPTION:
Study Description:

Between 10% and 15% of patients with endogenous hypercortisolism (Cushing syndrome) have ectopic (non-pituitary) production of adrenocorticotropin hormone (ACTH) that causes cortisol excess. In approximately 50% of these patients, the tumoral source of ACTH cannot be found initially despite very detailed and extensive imaging, including studies such as computed tomography, magnetic resonance imaging, and octreotide scan (Octreoscan) using the standard dose of indium- 111 pentetreotide ([111In-DTPA-D-Phe]-pentetreotide). The sensitivity and specificity of structurally based imaging studies depends on anatomic alterations and the size of the tumor. In contrast, positron emission tomography (PET) and somatostatin ligand imaging detect pathologic tissue based on physiologic and biochemical processes within the abnormal tissue.

This protocol tests the ability of [18F]-L-3,4-dihydroxyphenylalanine (18F-DOPA) PET, and the somatostatin imaging analogue, 68Ga-DOTATATE-PET, to localize the source of ectopic ACTH production.

Objectives:

Primary Objectives:

* To determine which imaging technique (F-DOPA PET/CT, 68Ga-DOTATATE PET/CT, standard CT, and/or standard MRI) has the best sensitivity.
* To determine if there is a combination of imaging tests with optimal diagnostic accuracy.

Secondary Objective:

-To evaluate a potential correlation between 18F-DOPA or 68Ga-DOTATATE uptake and the type of tumor, its size, SSTR expression or proliferative activity.

Exploratory Objectives:

* To evaluate the ability of gated cardiac imaging with CT and MRI to improve the detection of retrocardiac lung lesions.
* To determine whether PET scans at an interval of less than one year localize tumors.

Endpoints:

Primary Endpoint:

-Imaging results and pathology of resected tumors

Secondary Endpoints:

-18F-DOPA or 68Ga-DOTATATE imaging results, tumor pathology, tumor size, proliferative index and SSTR expression.

Exploratory Endpoints:

* Gated cardiac imaging CT and/or MRI; all other imaging results, tumor pathology.
* Imaging results and pathology of resected tumors.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* 18 - 90 years of age
* Medical history of ectopic Cushing syndrome or diagnosed with the possibility of ectopic Cushing syndrome
* For females of reproductive potential: agreement to use highly effective contraception for at least 2 weeks before any PET scan
* Ability of subject to understand and the willingness to sign a written informed consent document
* Stated willingness to comply with all study procedures and availability for the duration of the study

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation; the radiation associated with PET and CT scans may be harmful to a developing fetus. Likewise the ingestion of radionuclides in breast milk has an unknown risk to an infant.
* Evidence of severe active infection
* Clinically significantly impaired cardiovascular function, abnormal coagulation in the absence of medically-indicated treatment (PT and PTT elevated by 30% above the normal values), hematopoietic (hematocrit less than 30%, hemoglobin below 10 g/dl, white count below 3000 K/UL, and platelets below 100,000 K/mm^3), hepatic (liver enzymes elevated by 4-fold above normal values), or renal function (plasma creatinine level over 2.1).
* Based on the clinical judgment of the attending physician, other medical problems may prompt exclusion.
* Body weight over 136 kg, which is the limit for the tables used in the scanning areas.
* Combined blood withdrawal during the six weeks preceding the study greater than 450 ml.
* Subjects who previously underwent ten or more F-DOPA PET/CT scans and ten or more DOTATATE scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-02-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine which imaging technique (F-DOPA PET/CT, 68Ga-DOTATATE PET/CT, CT, and/or MRI) has the best sensitivity. | 6-12 months
  Subjects will be imaged every 6-12 months until tumor is found
To determine if there is a combination of imaging tests with optimal diagnostic accuracy. | 6-12 months
  subjects will be imaged every 6-12 months until tumor is found

SECONDARY OUTCOMES:
To evaluate a potential correlation between 18F-DOPA or 68Ga-DOTATATE uptake and the type of tumor, its size, SSTR expression or proliferative activity. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
On request, IPD related to a publication will be made available.
Supporting Information: CSR, Analytic Code
Time Frame: Start at the time of publication, for five years unless the study investigators leave NIH
Access Criteria: The PI will review requests and will provide data to investigators who wish to perform meta-analysis with other manuscript results. Data will be provided as an anonymized excel spread sheet.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-CH-0028.html